CLINICAL TRIAL: NCT04259073
Title: Does Pregabalin Improve Post-operative Pain After C-section Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital Universitaire Fattouma Bourguiba (Other)
Responsible Party: Principal Investigator, Khemili Malek, Principal investigator, Hôpital Universitaire Fattouma Bourguiba
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KMalek
Record Dates: First submitted 2020-02-03; First posted 2020-02-06 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Postoperative Pain
Keywords: postoperative pain; pregabalin; cesarean section
MeSH Terms: conditions — Pain, Postoperative | interventions — Pregabalin; Focal Adhesion Protein-Tyrosine Kinases; E1A-Associated p300 Protein

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group C (Placebo Comparator): two capsules filled with sugar
  Interventions: Drug: Placebos
- Group P150 (Active Comparator): two capsules; one of them containing sugar (like the placebo one), the other is the active drug (pregabalin 150 mg)
  Interventions: Drug: Pregabalin 150mg
- Group P300 (Active Comparator): two capsules of pregabalin (150 mg)
  Interventions: Drug: Pregabalin 300mg

INTERVENTIONS:
Drug: Pregabalin 150mg — two capsules, one is placebo, the other correspond to pregabalin 150 mg ingested orally one hour before cesarean section
  Other Names: P150
  Arms: Group P150
Drug: Placebos — two capsules filled with sugar ingested orally one hour before cesarean section
  Other Names: C
  Arms: Group C
Drug: Pregabalin 300mg — two capsules of pregabalin 150 mg ingested orally one hour before cesarean section
  Other Names: P300
  Arms: Group P300

SUMMARY:
Pregabalin due to its antihyperalgesic effect, has proven its efficacy on neuropathic pain, essentially in nociceptive surgeries. Few studies have attempted to identify the utility of pregabalin as a premedication before cesarean delivery.

The investigators aimed to determine whether or not pregabalin as premedication improves analgesia post cesarean delivery.

DETAILED DESCRIPTION:
The investigators conducted a controlled, randomised, prospective and double-blind trial. One hundred thirty eight participants were included, with American Society of Anesthesiologists physical status classification of I to II, with pregnancies of at least 36 weeks of gestation who were scheduled for elective caesarean delivery under spinal anaesthesia. One hour before induction of anaesthesia participants received a capsule containing sugar placebo (placebo group), pregabalin 150 mg or pregabalin 300 mg. Data related to surgical history, pre-existing medical problems, indications for cesarean and peroperative hemodynamic changes were analyzed. The primary outcome was first analgesic request. Secondary outcomes included maternal pain scores at rest and during movement, rescue analgesics consumption, sedation, nausea, vomiting, pruritus and Apgar scores. All maternal secondary outcome variables were recorded 0, 2, 4, 6, 12, 18, and 24 h after delivery. Common side effects linked to pregabalin such as somnolence, blurred or abnormal vision, or fetal distress were collected.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists class I or II
* single pregnancies at term
* under spinal anesthesia

Exclusion Criteria:

* conversion to general anesthesia
* post partum hemorrhage requiring specific resuscitation
* local anesthetic toxicity
* violation of the protocol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-10-10 (Actual)

PRIMARY OUTCOMES:
Time to first analgesic request | 24 hours
  in minutes, the time between the end of the operation to the first demand of analgesics

SECONDARY OUTCOMES:
Visual analog scale (VAS) at rest and movement | 24 hours
  Checked at hours 2, 4, 6,12,18 and 24 post operatively
Maternal satisfaction | 24 hours
  Measured by a Visual Analog Scale, ranging from 0 to 100; 0=not satisfied at all
Maternal consumption of paracetamol postoperatively | 24 hours
  grams
Apgar scores | 1 and 5 minutes after birth
  Ranging from 0 to 10; 7 to 10 correspond to an excellent condition
Heart rate | Per operative period
  beats per minute
Non-invasive blood pressure | Per operative period
  measured in millimeters of mercury
Visual disturbances | 24 hours post operatively
  present or not
Fluids administered to the mother per operatively | Per operative period
  in milliliters
Dose of ephedrine administered to the mother per operatively | Per operative period
  in milligrams
Ramsay score for sedation | 24 hours post operatively
  Ranging from 1 to 6

CONTACTS AND LOCATIONS:
Overall Officials: Malek Khemili, Resident, Principal Investigator — Fattouma Bourguiba Hospital ICU
Locations (1):
- Monastir maternity and neonatology center, Monastir, Tunisia

IPD SHARING:
Plan to Share IPD: Yes
principal outcomes measured in the study
Supporting Information: Study Protocol, SAP, CSR
Time Frame: March 2020 for one year
Access Criteria: after request by mailing

REFERENCES:
- [Background] El Kenany S, El Tahan MR. Effect of preoperative pregabalin on post-caesarean delivery analgesia: a dose-response study. Int J Obstet Anesth. 2016 May;26:24-31. doi: 10.1016/j.ijoa.2015.11.001. Epub 2015 Nov 12. PMID 26718698
- [Background] Felder L, Saccone G, Scuotto S, Monks DT, Carvalho JCA, Zullo F, Berghella V. Perioperative gabapentin and post cesarean pain control: A systematic review and meta-analysis of randomized controlled trials. Eur J Obstet Gynecol Reprod Biol. 2019 Feb;233:98-106. doi: 10.1016/j.ejogrb.2018.11.026. Epub 2018 Dec 12. PMID 30583095